CLINICAL TRIAL: NCT05409560
Title: Analysis of Core Temperature Afterdrop and Factors Associated With Afterdrop in Cold-water Swimming
Brief Title: Core Temperature Afterdrop in Cold-water Swimming
Acronym: THERMOCOLD
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: THERMOCOLD
Record Dates: First submitted 2022-04-17; First posted 2022-06-08 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2022-06

CONDITIONS: Hypothermia, Accidental; Cold Water Swimming
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cold water swimmers: swimmers participating in the 6-hour cold water swim, qualifying for the English Channel Swim
  Interventions: Other: Swimming participants in the 6-hour cold water swim

INTERVENTIONS:
Other: Swimming participants in the 6-hour cold water swim — The 6-hour cold water swim was the qualifying swim for the English Channel swim during the Channel Swim Camp Dinard 2021 and participants were the swimmers registered for the 6-hour cold water swim who volunteered to participate in this study

SUMMARY:
A significant risk associated with hypothermia during exercise in a cold environment is the core temperature (T°core) afterdrop, which corresponds to a continuous fall in T°core during rewarming after hypothermia. However, the rate and predictors of the afterdrop are unclear, particularly during prolonged cold water swimming.

The investigators propose to measure the changes in T°core during and after a cold water swim at 12.5-13°C qualifying for English Channel swim and to test the impact of anthropometric and swimming parameters on the duration of the T°core afterdrop. The hypotheses are that afterdrop is common during a prolonged cold water swimming event and that protective factors against T°core drop during cold water swimming (increased body fat and BMI) might, conversely, be associated with prolonged afterdrop.

ELIGIBILITY:
Inclusion Criteria:

* swimmers taking part in the Channel Swim Camp
* swimmers above 18 years of age
* swimmers willing and able to give informed consent for participation in the study

Exclusion Criteria:

* swallowing disorder
* chronic gastrointestinal disease
* MRI scheduled within 48 hours after the race.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Swimmers participating in the 6-hour cold-water swim, qualifying for the English Channel swim at the Channel Swim Camp (Dinard, France).
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Change in Body Core Temperature | Continuous measurement was collected from 30 minutes before the race until 2 hours after the end of the race for each swimmer
  Measurement of Body Core Temperature using an ingestible electronic sensor (e-Celsius®, BodyCap , Caen, France) which provide a continuous validated measurement

SECONDARY OUTCOMES:
Body composition, body mass | One measurement assessed the day before the race
  Fat mass (in kg, % of body mass [fat mass and body mass were combined to report % of body mass) was measured using bioelectrical impedance analysis (mBCA 525, Seca, Germany).
Body composition, fat-free mass | One measurement assessed the day before the race
  Fat-free mass (in kg, % of body mass [fat-free mass and body mass were combined to report % of body mass) was measured using bioelectrical impedance analysis (mBCA 525, Seca, Germany).
Body composition, muscle mass | One measurement assessed the day before the race
  Muscle mass (in kg, % of body mass [muscle mass and body mass were combined to report % of body mass) was measured using bioelectrical impedance analysis (mBCA 525, Seca, Germany).
Distance | The distance of swimming was collected from the organisers immediately after the race
  Distance of the swimming
Duration | The duration of swimming was collected from the organisers immediately after the race
  Duration of the swimming
Individual characteristics, gender | One evaluation assessed the day before the race
  The variable collected was the gender of participants
Individual characteristics, age | One evaluation assessed the day before the race
  The variables collected was the age of participants
Individual characteristics, swimming habits | One evaluation assessed the day before the race
  The variables collected was the swimming distance per week (total, swimming pool and open water)
Individual characteristics, training in cold environment | One evaluation assessed the day before the race
  The variable collected was the type of specific training in cold environment (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided